CLINICAL TRIAL: NCT01829711
Title: A Pivotal Multicenter Trial of Moxetumomab Pasudotox in Relapsed/ Refractory Hairy Cell Leukemia
Brief Title: Moxetumomab Pasudotox for Advanced Hairy Cell Leukemia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: MedImmune LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 130106; 13-C-0106 (Other: CTEP); CD-ON-CAT-8015-1053 (Other: MedImmune)
Record Dates: First submitted 2013-04-09; First posted 2013-04-11 (Estimated); Results first posted 2018-08-27 (Actual); Last update posted 2020-04-08 (Actual); Status verified 2020-03

CONDITIONS: Leukemia, Hairy Cell
Keywords: Moxetumomab Pasudotox; CAT-8015; Anti-cd22 recombinant immunotoxin; Biologic Therapy; Monoclonal Antibody; Pseudomonas Exotoxin; Targeted Therapy
MeSH Terms: conditions — Leukemia, Hairy Cell | interventions — immunotoxin HA22

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Moxetumomab pasudotox 40 µg/kg (Experimental): Patients will receive Moxetumomab Pasudotox intravenously (IV) over 30 minutes on days 1, 3, 5 of each 28 day cycle for a maximum of 6 cycles or until disease progression, unacceptable toxivity, initiation of alternate therapy or documented CR.
  Interventions: Drug: Moxetumomab pasudotox; Drug: IV Bag Protectant for Moxetumomab pasudotox

INTERVENTIONS:
Drug: Moxetumomab pasudotox
Drug: IV Bag Protectant for Moxetumomab pasudotox

SUMMARY:
Background:

- Moxetumomab pasudotox is an experimental non-chemotherapy cancer treatment drug. It targets CD22, a molecule on the surface of essentially all hairy cell leukemia cells. Moxetumomab pasudotox binds to CD22, goes into the cell, and releases a toxin which kills the cell. In a phase I trial it had activity in relapsed/refractory hairy cell leukemia with safety profile supporting further clinical study (http://ncbi.nlm.nih.gov/pubmed/22355053). This is a phase III multicenter trial designed to confirm these results.

DETAILED DESCRIPTION:
Background:

* Hairy cell leukemia (HCL) is an indolent B-cell leukemia comprising 2% of all leukemias, or approximately 900 of the 44,000 new cases of leukemia/year in the US
* Over the last two decades, immunotoxin research has accumulated to support a role for CD22-targeted therapy in the treatment of HCL.
* Moxetumomab pasudotox is a recombinant immunotoxin containing an Fv fragment of an anti-CD22 monoclonal antibody and truncated Pseudomonas exotoxin.
* Moxetumomab pasudotox has demonstrated a high complete response (CR) rate in patients with chemoresistant HCL and has shown activity in pediatric acute lymphoblastic leukemia as well.
* Modification of the structure of moxetumomab pasudotox has greatly improved binding and cytotoxicity toward CD22 expressing malignant cells compared to the precursor molecule. Preclinical and clinical studies have demonstrated that this increase in binding affinity results in improved antitumor activity and tolerability
* Currently there are no approved agents with significant efficacy for HCL patients after failure of standard therapy

Design:

* This is a multicenter, single-arm study of moxetumomab pasudotox in patients with relapsed/refractory hairy cell leukemia.
* 77 patients will be enrolled to receive moxetumomab pasudotox intravenously (IV) on days 1, 3 and 5 of each 28 day cycle for a maximum of 6 cycles or until disease progression, unacceptable toxicity occurs, the subject begins alternate therapy, or documented CR (for subjects who have no assessable minimal residual disease and not to exceed 6 cycles). If less than or equal to 2 of the first 25 patients do not achieve durable CR, no additional patients will be accrued.
* The overall IRB accrual ceiling is currently set at 80 to allow for a small number of patients that cannot be assessed for response.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Patients must have histologically confirmed hairy cell leukemia or hairy cell leukemia variant .with a need for therapy
* Patients must be Pseudomonas-immunotoxin naive
* Patients must have had at least 2 prior purine analogs, or at least 1 course of purine analog and 1 of either rituximab or BRAF inhibitor.
* Men or women age greater than or equal to 18 years.
* ECOG performance status less than or equal to 2.
* Patients must have adequate organ function

EXCLUSION CRITERIA

* Patients who have had chemotherapy, immunotherapy or radiotherapy within 4 weeks prior to entering the study.
* Patients who are receiving any other investigational agents.
* Patients with known brain metastases should be excluded from this clinical trial
* Patients with clinically significant ophthalmologic findings during screening
* Pregnant or breastfeeding females.
* Positive for Hepatitis B core antibody or surface antigen unless the patient is on Lamivudine or Entecavir and Hepatitis B Viral DNA load is less than 2000 IU/mL.
* Active second malignancy requiring treatment other than minor resection of indolent cancers like basal cell and squamous skin cancers
* HIV-positive patients unless taking appropriate anti-HIV medications with a CD4 count of greater than 200.
* History of allogeneic bone marrow transplant.
* Patients with history of both thromboembolism and known congenital hypercoagulable conditions.
* Uncontrolled pulmonary infection, pulmonary edema.
* Adequate oxygen saturation
* Radioimmunotherapy within 2 years prior to enrollment in study.
* Adequate hematologic function
* Adequate lung function
* Patients with history of thrombotic microangiopathy or thrombotic microangiopathy / hemolytic uremic syndrome
* Patients with QTc interval (Friderica) elevation > 500 msec based on at least 2 separate 12-lead ECGs
* Patient on high dose estrogen
* Patients with clinical evidence of disseminated intravascular coagulation

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2013-04-29 (Actual); Primary Completion 2017-05-24 (Actual); Study Completion 2019-04-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MedImmune LLC, Study Director — MedImmune LLC
Locations (34):
- United States (9):
  - Research Site, Duarte, California
  - Research Site, Los Angeles, California
  - Research Site, Miami, Florida
  - Research Site, Chicago, Illinois
  - Research Site, Baltimore, Maryland
  - Research Site, Bethesda, Maryland
  - Research Site, Albuquerque, New Mexico
  - Research Site, New York, New York
  - Research Site, Houston, Texas
- Belgium (2):
  - Research Site, Antwerp
  - Research Site, Ghent
- Research Site, Edmonton, Alberta, Canada
- Research Site, Brno, Czechia
- France (6):
  - Research Site, Caen
  - Research Site, Le Chesnay
  - Research Site, Pessac
  - Research Site, Pierre-Bénite
  - Research Site, Rouen
  - Research Site, Strasbourg
- Germany (3):
  - Research Site, Berlin
  - Research Site, Giessen
  - Research Site, Heidelberg
- Research Site, Dublin, Ireland
- Research Site, Haifa, Israel
- Italy (4):
  - Research Site, Bologna
  - Research Site, Genova
  - Research Site, Milan
  - Research Site, Siena
- Research Site, Bergen, Norway
- Poland (2):
  - Research Site, Gdansk
  - Research Site, Lodz
- Research Site, Belgrade, Serbia
- Research Site, Barcelona, Spain
- Research Site, Sutton, United Kingdom

REFERENCES:
- [Background] Bouroncle BA. Thirty-five years in the progress of hairy cell leukemia. Leuk Lymphoma. 1994;14 Suppl 1:1-12. PMID 7820038
- [Background] Jemal A, Siegel R, Ward E, Murray T, Xu J, Thun MJ. Cancer statistics, 2007. CA Cancer J Clin. 2007 Jan-Feb;57(1):43-66. doi: 10.3322/canjclin.57.1.43. PMID 17237035
- [Background] Sharpe RW, Bethel KJ. Hairy cell leukemia: diagnostic pathology. Hematol Oncol Clin North Am. 2006 Oct;20(5):1023-49. doi: 10.1016/j.hoc.2006.06.010. PMID 16990105
- [Background] Kreitman RJ, Tallman MS, Robak T, Coutre S, Wilson WH, Stetler-Stevenson M, Fitzgerald DJ, Lechleider R, Pastan I. Phase I trial of anti-CD22 recombinant immunotoxin moxetumomab pasudotox (CAT-8015 or HA22) in patients with hairy cell leukemia. J Clin Oncol. 2012 May 20;30(15):1822-8. doi: 10.1200/JCO.2011.38.1756. Epub 2012 Feb 21. PMID 22355053
- [Background] Kreitman RJ, Dearden C, Zinzani PL, Delgado J, Karlin L, Robak T, Gladstone DE, le Coutre P, Dietrich S, Gotic M, Larratt L, Offner F, Schiller G, Swords R, Bacon L, Bocchia M, Bouabdallah K, Breems DA, Cortelezzi A, Dinner S, Doubek M, Gjertsen BT, Gobbi M, Hellmann A, Lepretre S, Maloisel F, Ravandi F, Rousselot P, Rummel M, Siddiqi T, Tadmor T, Troussard X, Yi CA, Saglio G, Roboz GJ, Balic K, Standifer N, He P, Marshall S, Wilson W, Pastan I, Yao NS, Giles F. Moxetumomab pasudotox in relapsed/refractory hairy cell leukemia. Leukemia. 2018 Aug;32(8):1768-1777. doi: 10.1038/s41375-018-0210-1. Epub 2018 Jul 20. PMID 30030507
- [Derived] Kreitman RJ, Dearden C, Zinzani PL, Delgado J, Robak T, le Coutre PD, Gjertsen BT, Troussard X, Roboz GJ, Karlin L, Gladstone DE, Kuptsova-Clarkson N, Liu S, Patel P, Rotolo F, Mitry E, Pastan I, Giles F; Study 1053 investigators. Moxetumomab pasudotox in heavily pre-treated patients with relapsed/refractory hairy cell leukemia (HCL): long-term follow-up from the pivotal trial. J Hematol Oncol. 2021 Feb 24;14(1):35. doi: 10.1186/s13045-020-01004-y. PMID 33627164
- [Derived] Abou Dalle I, Ravandi F. Moxetumomab pasudotox for the treatment of relapsed and/or refractory hairy cell leukemia. Expert Rev Hematol. 2019 Sep;12(9):707-714. doi: 10.1080/17474086.2019.1643231. Epub 2019 Aug 1. PMID 31298972
- See also: NIH Clinical Center Detailed Web Page — http://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2013-C-0106.html
- See also: 130106_(CD-ON-CAT-8015-1053)_current_SAP_redacted_PDF-A — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=3161&filename=CD-ON-CAT-8015-1053_current_SAP_redacted_PDF-A.pdf
- See also: Protocol-cd-on-cat-8015-1053-amendment-9_redacted_PDF-A — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=3161&filename=protocol-cd-on-cat-8015-1053-amendment-9_redacted_PDF-A.pdf

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted across 14 countries (the USA, France, Italy, Germany, Belgium, Canada, Czech Republic, Ireland, Israel, Norway, Poland, Serbia, Spain, and United Kingdom).
Groups:
- Moxetumomab Pasudotox 40 µg/kg: Participants received intravenous infusion of moxetumomab pasudotox 40 µg/kg on Days 1, 3, and 5 of each 28-day cycle for up to 6 cycles, until documentation of complete response, progressive disease, initiation of alternate therapy, or unacceptable toxicity.
Period: Overall Study
Arm/Group | Moxetumomab Pasudotox 40 µg/kg
Started | 80
Completed | 37
Not Completed | 43
Not completed — Lost to Follow-up | 2
Not completed — Withdrawal by Subject | 3
Not completed — Death | 4
Not completed — Started new therapies | 17
Not completed — Adverse Event | 3
Not completed — Due to progression of disease | 13
Not completed — Due to lack of response | 1

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) population included participants who entered into the study and treated with moxetumomab pasudotox.
Arm/Group | Moxetumomab Pasudotox 40 µg/kg
Number analyzed (Participants) | 80
Age, Continuous [Mean (Standard Deviation); unit: Years] | 60.3 (11.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 63
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5
  Not Hispanic or Latino | 67
  Unknown or Not Reported | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 70
  More than one race | 0
  Unknown or Not Reported | 8

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Durable Complete Response (CR) Assessed by Blinded Independent Central Review
Description: Durable CR was defined as overall response that meets blood, bone marrow and imaging criteria for CR, followed by a >180 day duration of hematologic remission (HR). CR requires all of the following to be present: No evidence of leukemic cells in peripheral blood and/or by routine H/E staining of bone marrow; Resolution of any hepatomegaly, splenomegaly, and abnormal (>= 2 cm minimum length) lymphadenopathy by CT or MRI (maximum diameter of spleen should be either < 17 cm or have decreased by >25% from its baseline.); HR requires normal complete blood count (CBC) as exhibited by: Neutrophils >= 1.5 x 10^9/L, Platelets >= 100 x 10^9/L, and hemoglobin >= 11.0 g/dL without transfusions or growth factors for at least 4 weeks.
Time Frame: Full disease assessment (CBC, bone marrow and imaging) at end of treatment (EOT; up to 24 weeks) and post EOT Day 181; CBC monthly for 6 months post EOT, every 3 months post Day 181 for first 2 years and every 6 months thereafter (approximately 6 years)
Population: The ITT population included participants who entered into the study and treated with moxetumomab pasudotox.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Moxetumomab Pasudotox 40 µg/kg
Number analyzed (Participants) | 80
Percentage of participants | 36.3 [25.8 to 47.8]

2. Primary Outcome: Percentage of Participants With Durable CR by Investigator's Assessment
Description: Durable CR was defined as overall response that meets blood, bone marrow and imaging criteria for CR, followed by a >180 day duration of HR. CR requires all of the following to be present: No evidence of leukemic cells in peripheral blood and/or by routine H/E staining of bone marrow; Resolution of any hepatomegaly, splenomegaly, and abnormal (>= 2 cm minimum length) lymphadenopathy by CT or MRI (maximum diameter of spleen should be either < 17 cm or have decreased by >25% from its baseline.); HR requires normal complete blood count (CBC) as exhibited by: Neutrophils >= 1.5 x 10^9/L, Platelets >= 100 x 10^9/L, and hemoglobin >= 11.0 g/dL without transfusions or growth factors for at least 4 weeks.
Time Frame: as for outcome 1
Population: The ITT population included participants who entered into the study and treated with moxetumomab pasudotox.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Moxetumomab Pasudotox 40 µg/kg
Number analyzed (Participants) | 80
Percentage of participants | 48.8 [37.4 to 60.2]

3. Secondary Outcome: Percentage of Participants With Minimal Residual Disease (MRD) Positive or MRD Negative CR Assessed by Blinded Independent Central Review
Description: The MRD status by blinded independent review refers specifically to results of central pathologist read of bone marrow biopsy by immunohistochemistry.
  The CR with Positive or Negative MRD requires all of the following to be present:
  * No evidence of leukemic cells in the peripheral blood and/or by routine H/E staining of bone marrow. Minimal Residual Disease: CR with HCL evident in blood or in bone marrow biopsy by immunohistochemistry.
  * Resolution of any hepatomegaly, splenomegaly, and abnormal (>= 2 cm minimum length) lymphadenopathy by CT or MRI. Although a normal spleen size is not defined, the maximum diameter of the spleen should be either < 17 cm or have decreased by >25% from its baseline.
  * Normal CBC as exhibited by: Neutrophils >= 1.5 x 10^9/L, Platelets >= 100 x 10^9/L, and hemoglobin >= 11.0 g/dL without transfusions or growth factors for at least 4 weeks.
Time Frame: Prior to each treatment cycle, EOT (up to 24 weeks), monthly from the EOT assessment until the Day 181 assessment (only for CBC), at follow-up visits every 3 months for the next 24 months, and every 6 months thereafter (approximately 6 years)
Population: The ITT population included participants who entered into the study and treated with moxetumomab pasudotox.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Moxetumomab Pasudotox 40 µg/kg
Number analyzed (Participants) | 80
Percentage of participants
  MRD negative CR | 33.8 [23.6 to 45.2]
  MRD positive CR | 7.5 [2.8 to 15.6]

4. Secondary Outcome: Percentage of Participants With MRD Positive or MRD Negative CR by Investigator's Assessment
Description: The MRD status by investigator refers to results of investigator assessment of bone marrow biopsy or bone marrow aspirate by immunohistochemistry and/or flow cytometry.
  The CR with Positive or Negative MRD requires all of the following to be present:
  * No evidence of leukemic cells in the peripheral blood and/or by routine H/E staining of bone marrow. Minimal Residual Disease: CR with HCL evident in blood or marrow by flow cytometry.
  * Resolution of any hepatomegaly, splenomegaly, and abnormal (>= 2 cm minimum length) lymphadenopathy by CT or MRI. Although a normal spleen size is not defined, the maximum diameter of the spleen should be either < 17 cm or have decreased by >25% from its baseline.
  * Normal CBC as exhibited by: Neutrophils >= 1.5 x 10^9/L, Platelets >= 100 x 10^9/L, and hemoglobin >= 11.0 g/dL without transfusions or growth factors for at least 4 weeks.
Time Frame: Prior to each treatment cycle, end of treatment, and at follow-up visits every 3 months for the next 24 months and every 6 months thereafter (Approximately 6 years)
Population: The ITT population included participants who entered into the study and treated with moxetumomab pasudotox.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Moxetumomab Pasudotox 40 µg/kg
Number analyzed (Participants) | 80
Percentage of participants
  MRD negative CR | 32.5 [22.4 to 43.9]
  MRD positive CR | 7.5 [2.8 to 15.6]

5. Secondary Outcome: Time to CR Assessed by Blinded Independent Central Review
Description: Time to CR was defined as the time from the start of moxetumomab pasudotox administration to the first documentation of CR.
Time Frame: as for outcome 3
Population: The ITT population included participants who entered into the study and treated with moxetumomab pasudotox. Time to CR was evaluated for participants who achieved CR per independent central review.
Measure: Median (Full Range); unit: Months
Arm/Group | Moxetumomab Pasudotox 40 µg/kg
Number analyzed (Participants) | 80
Months | 5.9 [1.8 to 13.2]

6. Secondary Outcome: Duration of CR Assessed by Blinded Independent Central Review
Description: Duration of CR was defined as the duration from documentation of CR to the time of relapse from CR. Relapse from CR was defined as any CR criteria (blood counts, imaging or bone marrow) no longer consistent with CR. CR requires all of the following to be present: No evidence of leukemic cells in peripheral blood and/or by routine H/E staining of bone marrow; Resolution of any hepatomegaly, splenomegaly, and abnormal (>= 2 cm minimum length) lymphadenopathy by CT or MRI (maximum diameter of spleen should be either < 17 cm or have decreased by >25% from its baseline); normal CBC as exhibited by: Neutrophils >= 1.5 x 10^9/L, Platelets >= 100 x 10^9/L, and hemoglobin >= 11.0 g/dL without transfusions or growth factors for at least 4 weeks.
Time Frame: as for outcome 3
Population: The ITT population included participants who entered into the study and treated with moxetumomab pasudotox. Duration of CR was evaluated for participants who achieved CR per independent central review.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Moxetumomab Pasudotox 40 µg/kg
Number analyzed (Participants) | 80
Months | 62.8 [35.7 to 62.8]

7. Secondary Outcome: Duration of Hematologic Remission
Description: Duration of HR was defined as the duration from documentation of HR to the time of relapse. HR was defined as the blood counts required for CR as normal CBC as exhibited by: Neutrophils >= 1.5 x 10^9/L, Platelets >= 100 x 10^9/L, and hemoglobin >= 11.0 g/dL without transfusions or growth factors for at least 4 weeks.
  Duration of HR was censored on the date of the last hematologic assessment for participants who have no documented relapse based on blood count prior to data cutoff, dropout, or initiation of alternative anticancer therapy.
Time Frame: as for outcome 3
Population: The ITT population included participants who entered into the study and treated with moxetumomab pasudotox. Duration of HR was evaluated for participants who achieved HR.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Moxetumomab Pasudotox 40 µg/kg
Number analyzed (Participants) | 80
Months | 45.8 [25.9 to 71.5]

8. Secondary Outcome: Time to Hematologic Remission
Description: Time to HR was defined as the time from the start of moxetumomab pasudotox administration to the first documentation of HR. HR was defined as the blood counts required for CR as normal CBC as exhibited by: Neutrophils >= 1.5 x 10^9/L, Platelets >= 100 x 10^9/L, and hemoglobin >= 11.0 g/dL without transfusions or growth factors for at least 4 weeks.
Time Frame: as for outcome 3
Population: The ITT population included participants who entered into the study and treated with moxetumomab pasudotox. Time to HR was evaluated for participants in the ITT population who achieved HR.
Measure: Median (Full Range); unit: Months
Arm/Group | Moxetumomab Pasudotox 40 µg/kg
Number analyzed (Participants) | 80
Months | 1.1 [0.2 to 12.9]

9. Secondary Outcome: Percentage of Participants With Objective Response (OR) Assessed by Blinded Independent Central Review
Description: The OR was defined as number of participants with a best response of CR or PR. CR requires all of following to be present: No evidence of leukemic cells in peripheral blood and/or by routine H/E staining of bone marrow; Resolution of any hepatomegaly, splenomegaly, and abnormal (>=2 cm minimum length) lymphadenopathy by CT or MRI (maximum diameter of spleen should be either <17 cm or have decreased by >25% from its baseline); normal CBC (Neutrophils >=1.5 x 10^9/L, Platelets >=100 x 10^9/L, and hemoglobin >=11.0 g/dL) without transfusions or growth factors for at least 4 weeks. PR requires all of following for a period of at least 4 weeks: >=50% decrease or normalization (<5.0 x 10^9/L) in peripheral blood lymphocyte count and >=50% reduction in lymphadenopathy and in abnormal haepatosplenomegaly by CT or MRI from pre-treatment baseline value; normal CBC as mentioned above or 50% improvement in CBC values over baseline without transfusions or growth factors for at least 4 weeks.
Time Frame: as for outcome 3
Population: The ITT population included participants who entered into the study and treated with moxetumomab pasudotox.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Moxetumomab Pasudotox 40 µg/kg
Number analyzed (Participants) | 80
Percentage of participants | 75.0 [64.1 to 84.0]

10. Secondary Outcome: Percentage of Participants With Objective Response by Investigator's Assessment
Description: as for outcome 9
Time Frame: as for outcome 4
Population: The ITT population included participants who entered into the study and treated with moxetumomab pasudotox.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Moxetumomab Pasudotox 40 µg/kg
Number analyzed (Participants) | 80
Percentage of participants | 78.8 [68.2 to 87.1]

11. Secondary Outcome: Time to Objective Response Assessed by Blinded Independent Central Review
Description: Time to OR was defined as the time from the start of moxetumomab pasudotox administration to the first documentation of OR (CR or PR).
Time Frame: as for outcome 3
Population: The ITT population included participants who entered into the study and treated with moxetumomab pasudotox. Time to OR was evaluated for participants who achieved OR per independent central review.
Measure: Median (Full Range); unit: Months
Arm/Group | Moxetumomab Pasudotox 40 µg/kg
Number analyzed (Participants) | 80
Months | 5.7 [1.8 to 12.9]

12. Secondary Outcome: Duration of Objective Response Assessed by Blinded Independent Central Review
Description: Duration of OR was defined as the time from the first documentation of objective response (CR or PR) to the date of relapse.
  Duration of OR was censored on the date of last disease assessment or hematologic assessment for participants who have no documented relapse prior to data cut-off, dropout, or the initiation of alternative anticancer therapy.
Time Frame: as for outcome 3
Population: The ITT population included participants who entered into the study and treated with moxetumomab pasudotox. Duration of OR was evaluated for participants who achieved OR per independent central review.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Moxetumomab Pasudotox 40 µg/kg
Number analyzed (Participants) | 80
Months | 66.7 [25.4 to 66.7]

13. Secondary Outcome: Progression-free Survival (PFS) Assessed by Blinded Independent Central Review
Description: The PFS was defined as the time from the start of moxetumomab pasudotox administration to the earliest date of a disease assessment showing a progressive disease/relapse, earliest date of hematologic relapse or date of death, whichever was earlier. The PFS was censored on the date of last disease assessment or hematologic assessment for participants who are alive with no documented relapse or PD prior to data cut-off, dropout, or the initiation of alternative anticancer therapy.
Time Frame: as for outcome 3
Population: The ITT population included participants who entered into the study and treated with moxetumomab pasudotox.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Moxetumomab Pasudotox 40 µg/kg
Number analyzed (Participants) | 80
Months | 41.5 [28.1 to 71.7]

14. Secondary Outcome: Time to Treatment Failure (TTF) Assessed by Blinded Independent Central Review
Description: The TTF was defined as the time from the start of moxetumomab pasudotox administration to the date of the first of relapse, progressive disease, initiation of alternative anticancer therapy, or death due to disease or disease-related complication. The TTF was censored on the date of last disease assessment or hematologic assessment for participants who are alive with no documented relapse or PD prior to data cut-off, dropout, or the initiation of alternative anticancer therapy and also censored for death not accompanied by relapse.
Time Frame: as for outcome 3
Population: The ITT population included participants who entered into the study and treated with moxetumomab pasudotox.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Moxetumomab Pasudotox 40 µg/kg
Number analyzed (Participants) | 80
Months | 41.5 [28.1 to 71.7]

15. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs) and Treatment Emergent Serious Adverse Events (TESAEs)
Description: An Adverse Event (AE) is any unfavourable and unintended sign, symptoms, or diseases temporally associated with use of study drug, whether or not considered related to study drug. A serious adverse event (SAE) is an AE that results in death, initial or prolonged inpatient hospitalization, life-threatening, persistent or significant disability/incapacity, congenital anomaly/birth defect, or an important medical event. TEAEs and TESAEs are defined as AEs and SAEs present at baseline that worsened in intensity after administration of study drug, or events absent at baseline that emerged after administration of study drug.
Time Frame: From the start of study treatment (Day 1) through 4-6 weeks after last dose of Cycle 6 (28-day cycle) (approximately 7 months)
Population: Safety population included participants who received at least 1 dose of moxetumomab pasudotox.
Measure: Count of Participants; unit: Participants
Arm/Group | Moxetumomab Pasudotox 40 µg/kg
Number analyzed (Participants) | 80
Participants
  Any TEAEs | 79
  Any TESAEs | 28

16. Secondary Outcome: Number of Participants With Abnormal Clinical Laboratory Results Reported as TEAEs
Description: An abnormal laboratory finding which required an action or intervention by the investigator, or a finding judged by the investigator to represent a change beyond the range of normal physiologic fluctuation were reported as AEs. The TEAEs are defined as AEs present at baseline that worsened in intensity after administration of study drug, or events absent at baseline that emerged after administration of study drug, up to 30 days after the last dose of study drug (approximately 7 months).
Time Frame: as for outcome 15
Population: Safety population included participants who received at least 1 dose of moxetumomab pasudotox.
Measure: Count of Participants; unit: Participants
Arm/Group | Moxetumomab Pasudotox 40 µg/kg
Number analyzed (Participants) | 80
Participants
  Anaemia | 17
  Disseminated intravascular coagulation | 1
  Febrile neutropenia | 5
  Iron deficiency anaemia | 1
  Leukopenia | 2
  Lymphopenia | 1
  Neutropenia | 4
  Thrombocytopenia | 3
  Activated partial thromboplastin time prolonged | 1
  Lymphocyte count decreased | 16
  Lymphocyte count increased | 1
  Neutrophil count decreased | 6
  Platelet count decreased | 9
  White blood cell count decreased | 8
  Aspartate aminotransferase increased | 15
  Blood albumin decreased | 1
  Blood alkaline phosphatase increased | 4
  Blood bicarbonate decreased | 2
  Blood bilirubin increased | 5
  Blood creatinine increased | 9
  Blood triglycerides increased | 1
  Gamma-glutamyltransferase increased | 1
  Lipase increased | 2
  Hyperglycaemia | 8
  Hyperkalaemia | 6
  Hypermagnesaemia | 3
  Hypernatraemia | 4
  Hypertriglyceridaemia | 2
  Hypoalbuminaemia | 16
  Hypocalcaemia | 19
  Hypoglycaemia | 2
  Hypokalaemia | 13
  Hypomagnesaemia | 6
  Hyponatraemia | 9
  Haematuria | 6
  Haemoglobinuria | 2
  Proteinuria | 1

17. Secondary Outcome: Number of Participants With Abnormal Vital Signs Reported as TEAEs
Description: An abnormal vital signs that were judged by the investigator to be medically significant were reported as AEs. The TEAEs are defined as AEs present at baseline that worsened in intensity after administration of study drug, or events absent at baseline that emerged after administration of study drug, up to 30 days after the last dose of study drug (approximately 7 months).
Time Frame: as for outcome 15
Population: Safety population included participants who received at least 1 dose of moxetumomab pasudotox.
Measure: Count of Participants; unit: Participants
Arm/Group | Moxetumomab Pasudotox 40 µg/kg
Number analyzed (Participants) | 80
Participants
  Dyspnoea | 9
  Dyspnoea exertional | 3
  Hypertension | 12
  Hypotension | 6
  Pyrexia | 25

18. Secondary Outcome: Number of Participants With Abnormal Electrocardiogram (ECG) Reported as TEAEs
Description: An abnormal ECG findings that were judged by the investigator to be medically significant were reported as AEs. The TEAEs are defined as AEs present at baseline that worsened in intensity after administration of study drug, or events absent at baseline that emerged after administration of study drug, up to 30 days after the last dose of study drug (approximately 7 months).
Time Frame: as for outcome 15
Population: Safety population included participants who received at least 1 dose of moxetumomab pasudotox.
Measure: Count of Participants; unit: Participants
Arm/Group | Moxetumomab Pasudotox 40 µg/kg
Number analyzed (Participants) | 80
Participants
  Angina pectoris | 2
  Atrial fibrillation | 1
  Atrioventricular block first degree | 3
  Bundle branch block left | 1
  Left ventricular dysfunction | 1
  Palpitations | 1
  Pericardial effusion | 1
  Sinus bradycardia | 2
  Sinus tachycardia | 6
  Supraventricular tachycardia | 1
  Tachycardia | 1
  Ventricular arrhythmia | 1

19. Secondary Outcome: Time to Reach Maximum Observed Plasma Concentration (Tmax) of Moxetumomab Pasudotox
Description: The Tmax of moxetumomab pasudotox is reported.
Time Frame: Cycle 1 Day 1 (pre-dose; 5 mins and 3 hr post dose); Cycle 1 Day 5 (pre-dose; 5 mins, 1 hr, 3 hr, and 6 hrs post dose); and Cycle 2 Day 1 (pre-dose; 5 mins and 3 hr post dose)
Population: Pharmacokinetic (PK) population included all participants who received at least 1 dose of moxetumomab pasudotox and provided at least 1 baseline and post-baseline concentration-time data point.
Measure: Median (Full Range); unit: Hours
Arm/Group | Moxetumomab Pasudotox 40 µg/kg
Number analyzed (Participants) | 80
Hours
  Cycle 1 Day 1: number analyzed (Participants) | 75
  Cycle 1 Day 1 | 0.567 [0.433 to 1.30]
  Cycle 1 Day 5: number analyzed (Participants) | 71
  Cycle 1 Day 5 | 0.550 [0.417 to 2.45]
  Cycle 2 Day 1: number analyzed (Participants) | 69
  Cycle 2 Day 1 | 0.583 [0.500 to 1.75]

20. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) of Moxetumomab Pasudotox
Description: The Cmax of moxetumomab pasudotox is reported.
Time Frame: as for outcome 19
Population: The PK population included all participants who received at least 1 dose of moxetumomab pasudotox and provided at least 1 baseline and post-baseline concentration-time data point.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Moxetumomab Pasudotox 40 µg/kg
Number analyzed (Participants) | 80
ng/mL
  Cycle 1 Day 1: number analyzed (Participants) | 75
  Cycle 1 Day 1 | 192 (162)
  Cycle 1 Day 5: number analyzed (Participants) | 71
  Cycle 1 Day 5 | 435 (233)
  Cycle 2 Day 1: number analyzed (Participants) | 69
  Cycle 2 Day 1 | 379 (262)

21. Secondary Outcome: Time of Last (Tlast) Measurable Concentration of Moxetumomab Pasudotox
Description: The Tlast of moxetumomab pasudotox is reported.
Time Frame: as for outcome 19
Population: as for outcome 20
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Moxetumomab Pasudotox 40 µg/kg
Number analyzed (Participants) | 80
Hours
  Cycle 1 Day 1: number analyzed (Participants) | 75
  Cycle 1 Day 1 | 0.841 (0.866)
  Cycle 1 Day 5: number analyzed (Participants) | 71
  Cycle 1 Day 5 | 3.37 (2.38)
  Cycle 2 Day 1: number analyzed (Participants) | 69
  Cycle 2 Day 1 | 2.16 (1.43)

22. Secondary Outcome: Area Under the Plasma Concentration-time Curve From Time Zero to Time of the Last Quantifiable Concentration (AUC0-last) of Moxetumomab Pasudotox
Description: The AUC0-last of moxetumomab pasudotox is reported.
Time Frame: as for outcome 19
Population: as for outcome 20
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | Moxetumomab Pasudotox 40 µg/kg
Number analyzed (Participants) | 80
ng*hr/mL
  Cycle 1 Day 1: number analyzed (Participants) | 75
  Cycle 1 Day 1 | 120 (261)
  Cycle 1 Day 5: number analyzed (Participants) | 71
  Cycle 1 Day 5 | 820 (721)
  Cycle 2 Day 1: number analyzed (Participants) | 69
  Cycle 2 Day 1 | 626 (610)

23. Secondary Outcome: Area Under the Plasma Concentration-time Curve From Time Zero to 3 Hours (AUC0-3hr) Post End of Moxetumomab Pasudotox
Description: The AUC0-3hr of moxetumomab pasudotox is reported.
Time Frame: Cycle 1 Day 1 (pre-dose; 5 mins and 3 hr post dose); Cycle 1 Day 5 (pre-dose; 5 mins, 1 hr, and 3 hr post dose); and Cycle 2 Day 1 (pre-dose; 5 mins and 3 hr post dose)
Population: as for outcome 20
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | Moxetumomab Pasudotox 40 µg/kg
Number analyzed (Participants) | 80
ng*hr/mL
  Cycle 1 Day 1: number analyzed (Participants) | 6
  Cycle 1 Day 1 | 869 (200)
  Cycle 1 Day 5: number analyzed (Participants) | 54
  Cycle 1 Day 5 | 856 (370)
  Cycle 2 Day 1: number analyzed (Participants) | 37
  Cycle 2 Day 1 | 1030 (333)

24. Secondary Outcome: Area Under the Plasma Concentration-time Curve From Time Zero to Infinity (AUC0-inf) of Moxetumomab Pasudotox
Description: The AUC0-inf of moxetumomab pasudotox is reported.
Time Frame: as for outcome 19
Population: The PK population included all participants who received at least 1 dose of moxetumomab pasudotox and provided at least 1 baseline and post-baseline concentration-time data point. Data for Cycle 1 Day 1 was not reported as no evaluable participants for the calculation of the concerned parameters (ie., data were not sufficient).
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | Moxetumomab Pasudotox 40 µg/kg
Number analyzed (Participants) | 80
ng*hr/mL
  Cycle 1 Day 1: number analyzed (Participants) | 0
  Cycle 1 Day 5: number analyzed (Participants) | 49
  Cycle 1 Day 5 | 1300 (742)
  Cycle 2 Day 1: number analyzed (Participants) | 22
  Cycle 2 Day 1 | 1470 (541)

25. Secondary Outcome: Area Under the Plasma Concentration-time Curve Extrapolated (AUCExt) of Moxetumomab Pasudotox
Description: The AUCExt of moxetumomab pasudotox is reported.
Time Frame: as for outcome 19
Population: as for outcome 20
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | Moxetumomab Pasudotox 40 µg/kg
Number analyzed (Participants) | 80
ng*hr/mL
  Cycle 1 Day 1: number analyzed (Participants) | 6
  Cycle 1 Day 1 | 13.2 (3.04)
  Cycle 1 Day 5: number analyzed (Participants) | 49
  Cycle 1 Day 5 | 14.3 (5.72)
  Cycle 2 Day 1: number analyzed (Participants) | 22
  Cycle 2 Day 1 | 20.2 (7.62)

26. Secondary Outcome: Systemic Clearance (CL) of Moxetumomab Pasudotox
Description: The CL of moxetumomab pasudotox is reported.
Time Frame: as for outcome 19
Population: as for outcome 24
Measure: Mean (Standard Deviation); unit: mL/hr/kg
Arm/Group | Moxetumomab Pasudotox 40 µg/kg
Number analyzed (Participants) | 80
mL/hr/kg
  Cycle 1 Day 1: number analyzed (Participants) | 0
  Cycle 1 Day 5: number analyzed (Participants) | 49
  Cycle 1 Day 5 | 44.6 (30.5)
  Cycle 2 Day 1: number analyzed (Participants) | 22
  Cycle 2 Day 1 | 31.8 (13.7)

27. Secondary Outcome: Terminal Half Life (t1/2) of Moxetumomab Pasudotox
Description: The t1/2 of moxetumomab pasudotox is reported.
Time Frame: as for outcome 19
Population: as for outcome 24
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Moxetumomab Pasudotox 40 µg/kg
Number analyzed (Participants) | 80
Hours
  Cycle 1 Day 1: number analyzed (Participants) | 0
  Cycle 1 Day 5: number analyzed (Participants) | 49
  Cycle 1 Day 5 | 1.38 (0.632)
  Cycle 2 Day 1: number analyzed (Participants) | 22
  Cycle 2 Day 1 | 1.39 (0.351)

28. Secondary Outcome: Percentage of Participants With Positive Anti-drug Antibodies (ADA), Neutralizing Anti-drug Antibodies (nAb) and Specificity (CD22 and PE38) Positive to Moxetumomab Pasudotox
Description: Participants with ADA positive, nAb positive, cluster of differentiation 22 (CD22) positive of ADA positive/NAb positive, and pseudomonas exotoxin 38 (PE38) positive of ADA positive/NAb positive to moxetumomab pasudotox at any visit are reported.
Time Frame: Pre-infusion on Day 1 of Cycles 1, 2, 3, and 5; at the End of Treatment (4 to 6 weeks after the last dose; approximately 7 months)
Population: Safety population included participants who received at least 1 dose of moxetumomab pasudotox.
Measure: Number; unit: Percentage of Participants
Arm/Group | Moxetumomab Pasudotox 40 µg/kg
Number analyzed (Participants) | 80
Percentage of Participants
  ADA positive | 87.5
  ADA and NAb positive | 83.8
  Specificity CD22 positive of ADA+/NAb+ | 55.2
  Specificity PE38 positive of ADA+/NAb+ | 98.5

ADVERSE EVENTS:
Time Frame: For TEAEs and TESAEs: From the start of study treatment (Day 1) through 4-6 weeks after last dose of Cycle 6 (28-day cycle) (approximately 7 months) All-cause mortality data: From the start of study treatment (Day 1) through end of study (approximately 6 years)
Arm/Group | Moxetumomab Pasudotox 40 µg/kg
All-Cause Mortality (participants affected / at risk) | 4/80
Serious Adverse Events (participants affected / at risk) | 28/80
Other Adverse Events (participants affected / at risk) | 77/80
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Moxetumomab Pasudotox 40 µg/kg (N=80)
Febrile neutropenia (Blood and lymphatic system disorders) | 2 (3)
Haemolytic uraemic syndrome (Blood and lymphatic system disorders) | 6 (6)
Left ventricular dysfunction (Cardiac disorders) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Neutropenic colitis (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Fatigue (General disorders) | 1 (1)
Multiple organ dysfunction syndrome (General disorders) | 1 (1)
Pain (General disorders) | 1 (1)
Pyrexia (General disorders) | 5 (5)
Clostridium difficile colitis (Infections and infestations) | 1 (1)
Erysipelas (Infections and infestations) | 1 (1)
Infection (Infections and infestations) | 1 (1)
Lung infection (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Pneumonia fungal (Infections and infestations) | 1 (1)
Sepsis syndrome (Infections and infestations) | 1 (1)
Septic shock (Infections and infestations) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 2 (2)
Infusion related reaction (Injury, poisoning and procedural complications) | 2 (2)
Blood creatinine increased (Investigations) | 1 (1)
Haptoglobin decreased (Investigations) | 1 (1)
Neutrophil count decreased (Investigations) | 1 (1)
Platelet count decreased (Investigations) | 1 (1)
Weight increased (Investigations) | 1 (1)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 (1)
Glioblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Mental status changes (Psychiatric disorders) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1)
Haematuria (Renal and urinary disorders) | 1 (1)
Renal failure (Renal and urinary disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pharyngeal cyst (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1)
Capillary leak syndrome (Vascular disorders) | 4 (5)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Moxetumomab Pasudotox 40 µg/kg (N=80)
Anaemia (Blood and lymphatic system disorders) | 17 (41)
Neutropenia (Blood and lymphatic system disorders) | 4 (5)
Sinus tachycardia (Cardiac disorders) | 6 (6)
Cataract (Eye disorders) | 4 (4)
Dry eye (Eye disorders) | 6 (6)
Vision blurred (Eye disorders) | 7 (8)
Abdominal distension (Gastrointestinal disorders) | 10 (12)
Abdominal pain (Gastrointestinal disorders) | 7 (7)
Abdominal pain upper (Gastrointestinal disorders) | 4 (5)
Constipation (Gastrointestinal disorders) | 18 (21)
Diarrhoea (Gastrointestinal disorders) | 17 (20)
Dyspepsia (Gastrointestinal disorders) | 4 (5)
Flatulence (Gastrointestinal disorders) | 5 (5)
Nausea (Gastrointestinal disorders) | 28 (48)
Vomiting (Gastrointestinal disorders) | 14 (17)
Asthenia (General disorders) | 10 (30)
Chills (General disorders) | 15 (18)
Face oedema (General disorders) | 11 (16)
Fatigue (General disorders) | 26 (40)
Non-cardiac chest pain (General disorders) | 4 (4)
Oedema (General disorders) | 4 (5)
Oedema peripheral (General disorders) | 31 (47)
Peripheral swelling (General disorders) | 4 (5)
Pyrexia (General disorders) | 22 (35)
Nasopharyngitis (Infections and infestations) | 4 (4)
Rhinitis (Infections and infestations) | 4 (4)
Sinusitis (Infections and infestations) | 4 (4)
Upper respiratory tract infection (Infections and infestations) | 5 (5)
Infusion related reaction (Injury, poisoning and procedural complications) | 5 (6)
Alanine aminotransferase increased (Investigations) | 17 (43)
Aspartate aminotransferase increased (Investigations) | 15 (38)
Blood alkaline phosphatase increased (Investigations) | 4 (8)
Blood bilirubin increased (Investigations) | 5 (14)
Blood creatinine increased (Investigations) | 8 (15)
Haptoglobin decreased (Investigations) | 6 (6)
Lymphocyte count decreased (Investigations) | 16 (73)
Neutrophil count decreased (Investigations) | 5 (10)
Platelet count decreased (Investigations) | 9 (18)
Weight increased (Investigations) | 6 (7)
White blood cell count decreased (Investigations) | 8 (15)
Decreased appetite (Metabolism and nutrition disorders) | 11 (12)
Hyperglycaemia (Metabolism and nutrition disorders) | 8 (15)
Hyperkalaemia (Metabolism and nutrition disorders) | 6 (8)
Hypernatraemia (Metabolism and nutrition disorders) | 4 (5)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 16 (51)
Hypocalcaemia (Metabolism and nutrition disorders) | 19 (39)
Hypokalaemia (Metabolism and nutrition disorders) | 13 (22)
Hypomagnesaemia (Metabolism and nutrition disorders) | 6 (8)
Hyponatraemia (Metabolism and nutrition disorders) | 9 (17)
Hypophosphataemia (Metabolism and nutrition disorders) | 19 (47)
Arthralgia (Musculoskeletal and connective tissue disorders) | 13 (22)
Back pain (Musculoskeletal and connective tissue disorders) | 12 (12)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 4 (4)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 5 (7)
Myalgia (Musculoskeletal and connective tissue disorders) | 11 (16)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 12 (14)
Dizziness (Nervous system disorders) | 8 (12)
Dysgeusia (Nervous system disorders) | 5 (5)
Headache (Nervous system disorders) | 26 (37)
Paraesthesia (Nervous system disorders) | 7 (8)
Anxiety (Psychiatric disorders) | 9 (9)
Insomnia (Psychiatric disorders) | 8 (9)
Haematuria (Renal and urinary disorders) | 5 (5)
Cough (Respiratory, thoracic and mediastinal disorders) | 7 (8)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 8 (10)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 5 (5)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 6 (8)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 5 (6)
Pruritus (Skin and subcutaneous tissue disorders) | 6 (12)
Rash (Skin and subcutaneous tissue disorders) | 4 (4)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 4 (5)
Flushing (Vascular disorders) | 4 (4)
Hypertension (Vascular disorders) | 12 (38)
Hypotension (Vascular disorders) | 6 (8)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
MedImmune has 60 days to review results communications prior to public release and may delete information that compromises on-going studies or is considered proprietary. This restriction is not intended to compromise the objective scientific integrity of the manuscript, it being understood that results shall be published regardless of outcome.

DOCUMENTS (2):
  • Statistical Analysis Plan (2017-07-25): https://cdn.clinicaltrials.gov/large-docs/11/NCT01829711/SAP_000.pdf
  • Study Protocol (2017-03-29): https://cdn.clinicaltrials.gov/large-docs/11/NCT01829711/Prot_001.pdf